CLINICAL TRIAL: NCT06833320
Title: A Double-blind, Prospective, Randomized Trial of Propranolol for the Treatment of Postoperative Chylothorax After Open Cardiac Surgery
Brief Title: Propranolol Treatment for Postoperative Chylothorax
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: June Wu (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, June Wu, Associate Professor of Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAV5303
Record Dates: First submitted 2024-12-18; First posted 2025-02-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Chylothorax; Congenital Heart Disease; Open Heart Surgery; Chylothorax
MeSH Terms: conditions — Heart Defects, Congenital; Chylothorax | interventions — Propranolol; 2-Propanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to propranolol or placebo in a 1:1 ratio
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo suspension will only have Ora-Blend
  Interventions: Drug: Placebo
- Propranolol hydrochloride (Active Comparator): Subjects will be randomized to receive 2mg/kg/day. Propranolol will be administered orally, either as a tablet or as a solution, in equal divided doses three times a day.
  Interventions: Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Propranolol will be administered as tablets. Participants who are too young to swallow pills will be given propranolol solution.
  Other Names: Propranolol; 2-Propanol, 1-[(1-methylethyl)amino]-3-(1- naphthalenyloxy)-, hydrochloride
  Arms: Propranolol hydrochloride
Drug: Placebo — Placebo suspension will only have Ora-Blend Medication Flavoring and Suspension Vehicle
  Other Names: Ora-Blend
  Arms: Placebo

SUMMARY:
Postoperative chylothorax is a serious complication after open heart surgery for pediatric patients with congenital heart disease (CHD). While it was thought to be mechanical injury to the thoracic duct, recent research demonstrated that there are intrinsically abnormal lung lymphatics in CHD patients, and after open heart surgery, the fluid shifts that occur overwhelms these abnormal lung lymphatics. As a result, postoperative chylothorax occurs. Propranolol has been found to be helpful in resolving postoperative chylothorax very quickly (9 days) in a subset of postoperative chylothorax patients (60%). However, it is not known why some patients respond and some do not. The investigators hypothesize that propranolol is safe to use in this patient population, and that certain clinical factors will predict propranolol response, but more importantly, some clinical factors can be optimize to allow more patients with postoperative chylothorax to respond to and benefit from propranolol. In order to improve the understanding of how propranolol works and to maximize benefit to patients, the investigators propose to perform a prospective, randomized, double-blind clinical trial to learn how to best use propranolol in patients with postoperative chylothorax.

DETAILED DESCRIPTION:
This clinical trial will prospectively enroll eligible patients and randomize them to placebo or propranolol (1:1). This study will aim to enroll 50 patients, randomized to 25 placebo and 25 propranolol treatment. After patients have been consented, registered, and screened, they will be entered into the study. Participants will be randomized to placebo or propranolol in a 1:1 ratio. Randomization will be double-blinded, and each enrolled participant will be given a number and receive coded medication from the research pharmacy. Patients may undergo a screening MR lymphangiogram (MRL) prior to starting treatment. The criteria for an MRL will require that no additional sedation be given, and patient or parent/legal guardian consents to an MRL. Thus, only patients who are already sedated, or who will be able to undergo the MRL without sedation, and who opts in to the MRL will be eligible. Propranolol or placebo will be administered for 9 days after reaching the lowest effective goal dose not to exceed 2mg/kg/day, or maximum tolerated dose, after which the study groups will be unmasked.

Participants who have ≥80% reduction in volume of chylothorax drainage after 9 days of treatment and who received propranolol are identified as "responders". They will be taken off the study officially at this point as no more study interventions will be given. They will be tapered off of propranolol gradually as clinically indicated.

Participants who have ≥80% reduction in volume of chylothorax drainage but who received placebo will be the "natural history cohort". This will serve to demonstrate, as baseline, the percentage of participants who naturally resolve their chylothorax without intervention.

Patients who have <80% reduction in chylothorax drainage and who received propranolol, will be categorized as initial "non-responders". They will be officially taken off the study.

Participants who have <80% reduction in chylothorax drainage and who received placebo are considered a control group. They will be given propranolol for 9 days as a single-arm, open study and re-evaluated after a 9-day treatment. After 9 days at goal dosing, they will receive the same treatment as the responders and non-responders in the propranolol-treated group.

ELIGIBILITY:
Inclusion Criteria:

* ≥7 days and ≤18 years old at time of original cardiac surgery
* Congenital structural cardiac anomaly necessitating surgical correction. Examples include but are not limited to: ASD, VSD, single ventricles, HLHS, Tetralogy of Fallot, transposition of great vessels, AV canal, heart transplant
* developed high output postoperative chylothorax (≥10mL/kg/day), or
* persistent chylous drainage at any volume for ≥7 days after open heart surgery for a congenital cardiac defect
* ≥70% lymphocytes, or
* pleural triglyeride (TG) ≥ half of serum TG, or chylomicron positive

  * for patients with lower than normal serum lymphocyte count (agedependent), ≥60% lymphocytes in pleural fluids
* Must have measurable output (chylothorax output in mL)
* Any level of respiratory support (room air, supplemental oxygen, CPAP/BIPAP, ventilatory support)
* Any level of inpatient support (ICUs, step-down units, floor)
* Study participants can be on concomitant treatment for postoperative chylothorax started prior to study initiation
* Study participants can continue on on-going treatment for their primary cardiac other medical conditions
* Study participants can initiate new treatments for their primary cardiac or other medical conditions during trial period
* Adequate renal function
* Not on dialysis
* No hemodynamically unstable bradycardia
* No systolic hypotension not corrected by pressor support
* Not in 2nd or 3rd degree heart block
* No history of asthma
* A parent or a legal guardian must sign a written informed consent and HIPAA Form
* Patients will be required to also be enrolled in a related study (AAAQ6902) which collects chylothorax fluid for cell isolation and genetic analysis

Exclusion Criteria:

* Pregnancy
* Renal failure at time of enrollment
* Hypotension despite pressor support
* Unstable bradycardia without capacity for pacing
* History of asthma or chronic bronchodilator therapy
* Uncontrolled hypoglycemia or hyperglycemia as per investigators' judgment
* Study participant will be removed from study if they failed 2 consecutive attempts to initiate propranolol (>10% drop in BP/HR from age-adjusted normative range)
* Study participant experiences ≥ Grade 3 AE (SAE)

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Daily heart rates recorded in flow chart and 1 hour after each dose | 24 days
  Safety outcome
Daily blood pressures recorded in flow chart and 1 hour after each dose | 24 days
  Safety outcome
Daily glucose levels | 24 days
  Safety outcome
Expected and unexpected AEs, per patient | 24 days
  Safety outcome
Days with documented chest tube (# days), CXR | 24 days
  Will also measure the daily output (volume) in the chest tube(s)
Initial volume of fluid drained (mL, mL/kg/day) | Day 0
  The volume at the initial day of postoperative chylothorax diagnosis
Days hospitalized | 6 months
  The length of hospital stay, from post-surgery to discharge

SECONDARY OUTCOMES:
Thyroglobulin (TG) lymphocyte count | 24 days
  The TG count will be analyzed from the postoperative chylothorax fluid.
Pre-operative and post-operative echocardiogram anatomic findings for patients with 4-chamber hearts | Pre-operative and up to 24 days
  This outcome will be reported as the percent of patients with normal LV function, normal RV function, and normal pulmonary artery pressure.
Pre-operative and post-operative echocardiogram anatomic findings for patients with single ventricle (SV) physiology | Pre-operative and up to 24 days
  This outcome will be reported as the percent of patients with normal ventricular function and normal pulmonary artery pressure.
Percent of patients with Type 1 anatomy | Day 0
  Screening MR lymphangiogram: An optional imaging study to define lymphatic anatomy subtype
Percent of patients with Type 2 anatomy | Day 0
  Screening MR lymphangiogram: An optional imaging study to define lymphatic anatomy subtype
Percent of patients with Type 3 anatomy | Day 0
  Screening MR lymphangiogram: An optional imaging study to define lymphatic anatomy subtype
Percent of patients with Type 4 anatomy | Day 0
  Screening MR lymphangiogram: An optional imaging study to define lymphatic anatomy subtype
Serum albumin | 24 days
  to be extracted from clinical lab results, if available
White Blood Cell (WBC) count | 24 days
  to be extracted from clinical lab results, if available
C-Reactive Protein (CRP) | 24 days
  to be extracted from clinical lab results, if available
Immunoglobulin level | 24 days
  to be extracted from clinical lab results, if available
AT3 titer | 24 days
  to be extracted from clinical lab results, if available
Protein S titer | 24 days
  to be extracted from clinical lab results, if available
Protein C titer | 24 days
  to be extracted from clinical lab results, if available
Hours on bypass during CHD surgery | During surgery
  The amount of time the participant was on bypass during heart surgery
Triglyceride level in chylothorax fluid | 24 days
  Triglyceride levels will be measured

CONTACTS AND LOCATIONS:
Overall Officials: June Wu, MD, Principal Investigator — Columbia University Irving Medical Center/ New York Presbyterian hospital
Locations (1):
- Columbia University Irving Medical Center/NewYork-Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The aggregate data can be shared. The plan is not to share individual participant data to protect their privacy.

REFERENCES:
- See also: This study demonstrated the risk of developing postoperative chylothorax after open heart surgery, and that developing of this complication leads to prolonged hospitalization/ICU stay, need for mechanical ventilatory support, and death — https://pubmed.ncbi.nlm.nih.gov/28552079/
- See also: Postoperative chylothorax is associated with high resource utilization (prolonged hospitalization and mechanical ventilatory support). — https://pmc.ncbi.nlm.nih.gov/articles/PMC5594187/
- See also: postoperative chlyothorax is associated with increased hospital stay, costs, and mortality. — https://pubmed.ncbi.nlm.nih.gov/24246545/
- See also: A review on postoperative chylothorax and lymphatic leakage. — https://pmc.ncbi.nlm.nih.gov/articles/PMC5620321/
- See also: Our clinical study showing a subset of patients responded to propranolol with improved outcomes (shorter hospital stays, shorter days with chest tubes, less infection/thrombus risks). — https://pubmed.ncbi.nlm.nih.gov/34583843/